CLINICAL TRIAL: NCT06749028
Title: Evaluation of the Efficacy of Phospholipid-Bound Omega-3 Versus Omega-3 Alone in Patients With Hypertriglyceridemia: A Randomized Clinical Trial
Acronym: OMEGA-PHYT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación del Caribe para la Investigación Biomédica (Other)
Collaborators: Naturmega (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202401OMEGA-PHYT
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia;Fatty Acids, Omega-3;phospholipids, Omega-3
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Phospholipids

STUDY DESIGN:
Intervention Model Description: PICOT
  * Population:Adult patients ≥ 18 years old diagnosed with hypertriglyceridemia, defined as triglycerides >150 mg/dL.
  * Intervention: Omega-3 + phospholipids.
  * Comparator: Omega-3.
  * Outcome: Reduction in triglyceride levels and inflammatory markers, improvement in HOMA-IR index, and Omega Index.
  * Time:12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In addition to the parties commonly masked in this clinical trial(e.g., participants, investigators, and outcome assessors), other parties be masked include:
  1. Data Analysts: If feasible, data analysts will be blinded to the intervention groups during data analysis to reduce bias in interpreting results.
  2. Study Coordinators or Site Staff: Those responsible for enrolling participants or managing study logistics will be masked to intervention assignments to prevent unintentional influence on participant behavior.
  3. Pharmacists or Treatment Preparers: Pharmacists will be blinded to the allocation of active versus placebo treatments
  4. Regulatory Reviewers or Monitors: External reviewers or monitors who audit the study will be masked to treatment allocation to ensure unbiased oversight.
  5. Statistical Reviewers for Interim Analyses: the statisticians conducting these will be masked to group allocations to preserve trial integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B: Comparator Arm: Omega-3 alone. (Active Comparator): Comparator Arm: Omega-3 alone
  Interventions: Dietary Supplement: Comparator Arm: Omega-3 alone.
- Group A: Intervention Arm: Omega-3 + Phospholipids. (Experimental): Intervention Arm: Omega-3 + Phospholipids.
  Interventions: Dietary Supplement: Intervention Arm: Omega-3 + Phospholipids.

INTERVENTIONS:
Dietary Supplement: Intervention Arm: Omega-3 + Phospholipids. — Intervention Arm: Omega-3 + Phospholipids.
  Arms: Group A: Intervention Arm: Omega-3 + Phospholipids.
Dietary Supplement: Comparator Arm: Omega-3 alone. — Comparator Arm: Omega-3 alone.
  Arms: Group B: Comparator Arm: Omega-3 alone.

SUMMARY:
Hypertriglyceridemia is a significant risk factor for cardiovascular diseases. Omega-3 fatty acids have been shown to reduce triglyceride levels, and their combination with phospholipids could offer additional benefits in improving lipid profiles and inflammatory markers. This study aims to evaluate the efficacy of combining omega-3 with phospholipids compared to omega-3 alone in patients with hypertriglyceridemia. The objective of the clinical trial is to provide robust evidence on the benefits of this combination in improving lipid profiles and reducing inflammation, which could have a significant impact on clinical practices and future dietary recommendations.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of combining omega-3 with phospholipids compared to omega-3 alone in patients with hypertriglyceridemia. The objective of the clinical trial is to provide robust evidence of the benefits of this combination in improving lipid profiles and reducing inflammation, which could significantly impact clinical practices and future dietary recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 to 65 years.
* Triglyceride levels ≥ 150 mg/dL and ≤ 500 mg/dL.
* Signed informed consent.

Exclusion Criteria:

* Use of omega-3 supplements in the last 3 months.
* Use of any lipid-lowering medication.
* Known allergy to the components of the treatment.
* Uncontrolled chronic diseases (e.g., renal failure, liver disease).
* Any type of cancer.
* Undergoing treatment for HIV.
* Pregnancy or breastfeeding.
* Use of substances or prescribed medications that may increase triglyceride levels (e.g., estrogens, atypical antipsychotics, etc.). -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Triglyceride Levels | 12 weeks
  Description: Evaluate the change in triglyceride levels (mg/dL) from baseline to 12 weeks.

SECONDARY OUTCOMES:
Reduction in Inflammatory Markers | 12 weeks
  Assess changes in levels of inflammatory markers such as High Sensivity CRP (C-reactive protein) and IL-6 (interleukin-6) from baseline to 12 weeks.
Improvement in HOMA-IR Index | 12 weeks
  Measure changes in the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) from baseline to 12 weeks.
Improvement in Omega Index | 12 weeks
  Assess changes in the Omega Index (percentage of omega-3 fatty acids in red blood cell membranes) from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Urina, PhD, Principal Investigator — Fundacion del Caribe para la investigación Biomedica
Locations (1):
- Fundacion del Caribe para la Investigación Biomedica, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: Yes
1. Purpose of Data Sharing: Explain why the personal data will be shared, such as to foster collaboration on additional research, validate results, or conduct broader analyses.
  2. Types of Data to be Shared: Describe the types of personal or sensitive data that will be shared, ensuring that only the necessary data for research will be provided.
  3. Confidentiality and Security Measures: Detail how personal data will be protected to ensure the privacy and confidentiality of participants. This could include anonymizing or pseudonymizing the data, using secure platforms for data exchange, and complying with legal regulations such as the General Data Protection Regulation (GDPR).
  4. Requirements for Researchers Receiving the Data: Specify the requirements for researchers receiving the data, such as signing confidentiality agreements and committing to use the data solely for the agre
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months
Access Criteria: 1. Who Will Have Access:
     * Principal Investigators (PIs) and Research Team
     * Collaborating Researchers
     * Regulatory Authorities
  2. What They Will Be Able to Access:
     Personal Data Study Data Supporting Information
  3. How They Will Be Able to Access It:
  Secure Data Platforms Access Request Process Data Access Agreements Anonymized or De-identified Data